CLINICAL TRIAL: NCT04567121
Title: Internet Technology Based Life-style and Care Intervention for Risk Factors of Non Communicable Diseases（NCD）-a Randomized, Controlled Trial in Communities Following Up for 50 Years
Brief Title: Internet Technology Based Life-style and Care Intervention for Risk Factors of Non Communicable Diseases（NCD）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20281-0-01
Record Dates: First submitted 2020-09-07; First posted 2020-09-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-05

CONDITIONS: Lifestyle Intervention; Non Communicable Diseases
Keywords: Internet Technology; lifestyle intervention; Non Communicable Diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive intervention group (Other): intensive life-style and care intervention
  Interventions: Behavioral: Intensive intervention group
- Standard intervention group (Other): standard life-style and care intervention
  Interventions: Behavioral: standard intervention group

INTERVENTIONS:
Behavioral: Intensive intervention group — Establish a team of chronic disease prevention managers (5 people), with each educator responsible for the intervention of 200 people. For sub-health population and chronic disease patients, there would be conducted health education interview twice, 4 calls, online communication 50 times once a year, controlling risk factors and making treatment plan.
  Arms: Intensive intervention group
Behavioral: standard intervention group — Conduct general health education without active management
  Arms: Standard intervention group

SUMMARY:
This study aims to control risk factors of non communicable diseases by life style and care intervention based on internet technology, looking forward to improve cardiovascular and cerebrovascular complications, diabetes and all-cause death.

DETAILED DESCRIPTION:
Cardiovascular and cerebrovascular diseases, diabetes, chronic obstructive pulmonary disease and malignant tumors are the main chronic diseases, which have been the most important cause of human death, consuming most health resources. In China, patients with cardiovascular and cerebrovascular diseases account for more than 40% of all causes of death. After half a century of research, we have a thorough understanding of risk factors of cardiovascular disease, including genetics, aging, ethnicity, physical activity decreases, unbalanced nutrition and calorie intake, smoking, obesity, hypertension, dyslipidemia, and glucose abnormalities, etc. Many factors can be corrected through health education, indicating that the occurrence of chronic diseases can be prevented through lifestyle changes and the control of risk factors.

This project collects risk factors of cardiovascular disease and establishes a real and reliable health database by conducting a cross-sectional survey of chronic diseases among residents of Tian Tong Yuan District (there are hundreds of thousands of people).On this basis, community health management network was established with internet technology. Meanwhile, prospective, open, community randomized and controlled lifestyle intervention studies were carried out. Intervention was conducted on risk factors of cardiovascular and cerebrovascular diseases, such as smoking, obesity, hypertension, lipid metabolism disorder, and hyperglycemia. For patients with chronic diseases, lifestyle intervention and health education should be carried out to improve the diagnosis rate and control rate. The project focuses on the impact of lifestyle interventions and health education on risk factor control, cardiovascular and cerebrovascular complications, diabetes and all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 25 years of age with two or more risk factors as follows, BMI≥24 or BMI≤18.5 kg/m2, smoking, active exercise less than 30 minutes every day, blood pressure higher than 130/85 mmHg, dyslipidemia, fasting glucose higher than 6.1mmol/l, fatty liver.
* Patients with hypertension, diabetes and ASCVD

Exclusion Criteria:

* Patients had not signed the consent form
* Patients with severe heart failure, hepatic failure, renal failure and malignant tumor.
* Patients planing pregnancy

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2070-01-01 (Estimated); Study Completion 2070-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence rate of new noncommunicable diseases | 2 year
  incidence rate of new noncommunicable diseases, for example, ASCVD, diabetes mellitus, hypertension
incidence rate of major adverse cardiovascular events | 2 years
  incidence rate of major adverse cardiovascular events, including nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
incidence rate of all-cause mortality | 2 years
  incidence rate of all-cause mortality in the population

SECONDARY OUTCOMES:
score of quality of life (SF-36 scale) | 2 years
  the improvement of quality of life
Reduce the economic burden on health | 2 years
  survey of health economic burden, calculate medical expenses

CONTACTS AND LOCATIONS:
Overall Officials: jianzhong xiao, PHD, Study Director — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No